CLINICAL TRIAL: NCT00864760
Title: A Relative Bioavailability Study of 800 mg Gabapentin Tablets Versus 400 mg Gabapentin Capsules Under Fasting Conditions
Brief Title: A Relative Bioavailability Study of Gabapentin 800 mg Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Responsible Party: Meena Venugopal, Director, Clinical R&D, Actavis Inc
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: P99-228
Record Dates: First submitted 2009-03-17; First posted 2009-03-19 (Estimated); Last update posted 2010-08-17 (Estimated); Status verified 2010-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Gabapentin; Healthy subjects
MeSH Terms: interventions — Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Gabapentin 800 mg tablets, single dose (1 tablet)
  Interventions: Drug: Gabapentin 800 mg tablets, single dose (1 tablet)
- B (Active Comparator): NEURONTIN® 400 mg capsules, single dose (2 capsules)
  Interventions: Drug: NEURONTIN® 400 mg capsules, single dose (2 capsules)

INTERVENTIONS:
Drug: Gabapentin 800 mg tablets, single dose (1 tablet) — A: Experimental Subjects received Purepac formulated products under fasting conditions
  Arms: A
Drug: NEURONTIN® 400 mg capsules, single dose (2 capsules) — B: Active comparator Subjects received Parke-Davis formulated products under fasting conditions
  Other Names: Gabapentin
  Arms: B

SUMMARY:
The purpose of this study is to compare the relative bioavailability of 800 mg Gabapentin Tablets by Purepac Pharmaceutical Co. with that of 400 mg (2 x 400 mg) NEURONTIN® by Parke-Davis under fasting conditions.

DETAILED DESCRIPTION:
Study Type: Interventional Study Design: Randomized, single-dose, two-way crossover design under fasting conditions

Official Title: A Relative Bioavailability Study of 800 mg Gabapentin Tablets versus 400 mg Gabapentin Capsules Under Fasting Conditions

Further study details as provided by Actavis Elizabeth LLC:

Primary Outcome Measures:

Rate and Extend of Absorption

ELIGIBILITY:
Inclusion Criteria:

* Screening Demographics: All volunteers selected for this study will be healthy men 18 to 45 years of age, inclusive, at the time of dosing. The weight range will not exceed ± 15% for height and body frame as per Desirable Weights for Men• 1983 Metropolitan Height and Weight Table.
* Screening Procedures: Each volunteer will complete the screening process within 28 days prior to Period I dosing. Consent documents for both the screening evaluation and HIV antibody determination will be reviewed, discussed, and signed by each potential participant before full implementation of screening procedures.
* Screening will include general observations, physical examination, demographics, medical and medication history, an electrocardiogram, sitting blood pressure and heart rate, respiratory rate and temperature. The physical examination will include, but may not be limited to, an evaluation of the cardiovascular, gastrointestinal, respiratory and central nervous systems.
* The screening clinical laboratory procedures will include:

  * HEMATOLOGY: hematocrit, hemoglobin, WBC count with differential, RBC count, platelet count
  * CLINICAL CHEMISTRY: serum creatinine, BUN, glucose, AST(GOT), ALT(GPT), albumin, total bilirubin, total protein, and alkaline phosphatase
  * HIV antibody and hepatitis B surface antigen screen
  * URINALYSIS: pH, albumin, sugar, acetone, bilirubin, occult blood and microscopic analysis
  * URINE DRUG SCREEN: ethyl alcohol. amphetamines. barbiturates, benzodiazepines, cannabinoids. cocaine metabolites, opiates and phencyclidine.

Exclusion Criteria:

* Volunteers with a recent history of drug or alcohol addiction or abuse.
* Volunteers with the presence ofa clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, immunologic, hematologic, endocrine, or neurologic system(s) or psychiatric disease (as determined by the medical investigator).
* Volunteers whose clinical laboratory test values are outside the accepted reference range and when confirmed on re-examination are deemed to be clinically significant.
* Volunteers demonstrating a positive hepatitis B surface antigen screen or a reactive HIV antibody screen.
* Volunteers demonstrating a positive drug abuse screen when screened for this study.
* Volunteers with a history of allergic response(s) to gabapentin or related drugs.
* Volunteers with a history of clinically significant allergies including drug allergies.
* Volunteers with a clinically significant illness during the 4 weeks prior to Period I dosing (as determined by the medical investigator.
* Volunteers who currently use tobacco products.
* Volunteers who have taken any drug known to induce or inhibit hepatic drug metabolism in the 30 days prior to Period I dosing.
* Volunteers who report donating greater than 150 mL of blood within 30 days prior to Period I dosing. All subjects will be advised not to donate blood for four weeks after completing the study.
* Volunteers who have donated plasma (e.g. plasmaphoresis) within 14 days prior to Period I dosing. All subjects will be advised not to donate plasma for four weeks after completing the study.
* Volunteers who report receiving any investigational drug within 30 days prior to Period I dosing.
* Volunteers who report taking any systemic prescription medication in the 14 days prior to Period I dosing.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 1999-06; Primary Completion 1999-06 (Actual); Study Completion 1999-06 (Actual)

PRIMARY OUTCOMES:
Rate and Extend of Absorption | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: James D. Carlson,, Pharm. D., Principal Investigator — PRACS Institute, Ltd.
Locations (1):
- PRACS Institute, Ltd., Fargo, North Dakota, United States